CLINICAL TRIAL: NCT05257330
Title: Evaluation of Non-Compressive Myelopathy in a Sample of Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdel-Ghaffar Ismail Fayed, Lecturer in Neurology, Al-Azhar University
Other Study IDs: 0000044
Record Dates: First submitted 2022-02-17; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Myelopathy; Non-Compressive
MeSH Terms: conditions — Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CSF Examination — Lumbar puncture for CSF Examination

SUMMARY:
An observational study will be conducted in the Department of Neurology at AlAzhar University Hospitals To study the etiological factors of non-compressive myelopathy in a sample of Egyptian patients

DETAILED DESCRIPTION:
Myelopathy is a collective term referring to any pathologic condition or neurologic deficit related to the spinal cord. Myelopathies are a frequent and potentially disabling neurologic emergency.(Sarbu et al., 2019).

Diseases of the spinal cord often have devastating consequences and imaging studies are indispensable for their diagnosis. The diagnostic approach must be based on the clinical context, the time elapsed since the onset of symptoms and signs, and the imaging findings (Herrera et al., 2020).

Myelopathies may be compressive or non-compressive, regarding to subarachnoid space obstruction (Kundu et al., 2018).

Noncompressive myelopathy (NCM) is described as "spinal cord involvement without detectable clinical and radiological evidence of spinal cord compression causing neurological deficit (Thangaraj et al., 2019).

There have been a few studies that have investigated Noncompressive myelopathy (NCM) in Africa as part of nontraumatic myelopathy. With very few studies focusing on NMOSD, Most of them focus on extrinsic compression and infectious diseases as important causes of myelopathy (Musubire et al., 2021) Comprehensive data on Egyptian patients with Non-compressive myelopathy (NCM) in the light of newer diagnostic criteria and serological tests are lacking. No study has been conducted to study the clinico-radiological profile of Non-compressive myelopathy (NCM) so far. In this study, we are putting an effort to convey our experience on etiological pattern of Non-compressive myelopathy (NCM) with special reference to its radiological features.

ELIGIBILITY:
Inclusion Criteria:

- Patients with acute, subacute, or chronic neurologic dysfunction (motor and sensory deficit, sphincteric involvement, and a well-defined upper sensory segmental level) consistent with myelopathy (with or without coexisting encephalopathy, neuropathy, or radiculopathy).

Exclusion Criteria:

* 1) Patients of myelopathy who did not undergo magnetic resonance imaging (MRI) of the spinal cord. 2) Spinal cord compression on MRI explaining patient's neurologic dysfunction. 3) History of previous trauma, acute coma and patients with definite cerebral symptoms incompatible with spinal pathology (e.g., aphasia, hemianopia, neglect, facial involvement). 4) Motor neuron disease (MND) 5)Degenerative ataxias.

Ages: 2 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute, subacute, or chronic neurologic dysfunction consistent with myelopathy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
To study the etiological factors of non-compressive myelopathy in a sample of Egyptian patients | 6 months
  study the clinico-radiological profile of Non-compressive myelopathy

CONTACTS AND LOCATIONS:
Overall Officials: Mohie-eldin T Mohamed, Professor, Principal Investigator — Al-Azhar Faculty of medicine
Locations (1):
- Al-Hussein and Sayed Galal Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
To study the etiological factors of Non-compressive Myelopathy in a sample of Egyptian patients